CLINICAL TRIAL: NCT05957081
Title: A Phase 1a/1b, First-in-Human, Open Label Study to Assess the Safety, Tolerability, and Pharmacokinetics of PMC-309 (Anti-VISTA), as Monotherapy and Combined With Pembrolizumab, in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study to Assess the Safety, Tolerability, and Blood Concentration of PMC-309
Acronym: MarkV-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAbcine (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarkV-01; KEYNOTE-E80 (Other: Merck Sharp & Dohme Corp); MK-3475-E80 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2023-05-26; First posted 2023-07-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: PMC-309 and Anti-VISTA
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 a: Part A: PMC-309 Monotherapy Dose Escalation (Experimental): Phase 1a will enroll participants with advanced or metastatic solid tumors to assess safety, tolerability, PK and clinical efficacy in response to treatment with PMC-309 as a monotherapy
  Dosage form and Route of administration: The duration of a treatment cycle is 3 weeks/21 days. Participants will be administered a weekly dose of PMC-309 per cycle as follows:
  * Cycle Week 1/Day 1
  * Cycle Week 2/Day 8 ± 2 days
  * Cycle Week 3/Day 15 ± 2 days PMC-309 will be administered intravenously over 1 hour (± 0.5 hours), after which participants will be observed for a period of 1.5 hours post administration.
  Interventions: Drug: PMC-309 monotherapy
- Phase 1a: Part B: PMC-309 Dose Escalation in Combination with Pembrolizumab (Experimental): Part B will establish the MTD/preliminary RP2D of PMC-309 when administered in combination with 200 mg pembrolizumab. Part B will be conducted after completion of Part A (PMC-309 monotherapy dose escalation) and before the commencement of Phase 1b.
  Dosage form and Route of administration: The duration of a treatment cycle is 3 weeks/21 days. Participants will be administered a weekly dose of PMC-309 plus one dose of pembrolizumab at 200 mg per cycle as follows:
  * Cycle Week 1/Day 1: pembrolizumab (administered first), followed by administration of PMC-309.
  * Cycle Week 2/Day 8 ± 2 days: PMC-309 only
  * Cycle Week 3/Day 15 ± 2 days: PMC-309 only. Both PMC-309 and pembrolizumab will be administered intravenously.
  Interventions: Drug: PMC-309 Dose Escalation in Combination with Pembrolizumab(KEYTRUDA®)
- Phase 1b: Dose Expansion (Experimental): Phase 1b will enroll participants after completion of DLT assessments for Phase 1a.
  Phase 1b will enroll participants with advanced or metastatic tumor types into 1 of 2 cohorts to assess response of monotherapy of PMC-309 and response of PMC-309 in combination with pembrolizumab.
  * Cohort A: PMC-309 monotherapy therapy
    - PMC-309 dosing will be at the preliminary RP2D, as identified in Phase 1a: Part A
  * Cohort B: PMC-309 plus pembrolizumab combination therapy - PMC-309 dosing will be as identified in Phase 1a: Part B in combination with 200 mg pembrolizumab Participants will be randomly assigned to Cohort A or Cohort B until 20 participants are enrolled in each cohort.
  Interventions: Drug: PMC-309 Dose Expansion

INTERVENTIONS:
Drug: PMC-309 monotherapy — PMC-309 will be administered intravenously.
  Other Names: Monotherapy
  Arms: Phase 1 a: Part A: PMC-309 Monotherapy Dose Escalation
Drug: PMC-309 Dose Escalation in Combination with Pembrolizumab(KEYTRUDA®) — Both PMC-309 and pembrolizumab will be administered intravenously. At the time of the combination therapy (Week 1/Day 1 of each cycle), participants will be dosed with pembrolizumab(KEYTRUDA®) first, administered over 0.5 hours (± 10 minutes). Following an interval of 1 hour (± 15 minutes), participants will be dosed with PMC-309 administered over 1 hour (± 0.5 hours), after which participants will be observed for a period of 1.5 hours post administration.
  Other Names: Combination Therapy
  Arms: Phase 1a: Part B: PMC-309 Dose Escalation in Combination with Pembrolizumab
Drug: PMC-309 Dose Expansion — Phase 1b will enroll participants with advanced or metastatic tumor types into 1 of 2 cohorts:
  * Cohort A: PMC-309 monotherapy therapy
    - PMC-309 dosing will be at the preliminary RP2D, as identified in Phase 1a: Part A
  * Cohort B: PMC-309 plus pembrolizumab(KEYTRUDA®) combination therapy - PMC-309 dosing will be as identified in Phase 1a: Part B in combination with 200 mg pembrolizumab(KEYTRUDA®)
  Other Names: Mono and Combination therapy
  Arms: Phase 1b: Dose Expansion

SUMMARY:
This is a Phase 1a/1b, first-in-human (FIH), open label study to evaluate the safety, tolerability, and pharmacokinetics (PK) of PMC-309, a mAb against the human VISTA ligand, in participants with advanced or metastatic solid tumors administered as a monotherapy and in combination with pembrolizumab.

DETAILED DESCRIPTION:
Phase 1a is a 2-part dose escalation; both part will adopt the modified toxicity probability interval (mTPI) design with a dose limiting toxicity (DLT) rate of 30% for dose finding.

* Part A is planned as a PMC-309 dose escalation.
* Part B: is planned as a PMC-309 dose escalation in combination with pembrolizumab.

Phase 1b is planned as a cohort expansion with PMC-309 administered as a monotherapy (Cohort A) at the preliminary recommended Phase 2 dose (RP2D) found at Phase 1a (Part A) and in combination with pembrolizumab (Cohort B) with PMC-309 at the maximum tolerated dose (MTD)/preliminary recommended Phase 2 dose (RP2D) found at Phase 1a (Part B).

A minimum of 67 participants are to be enrolled to the study.

Treatment Groups: Phase 1a Part A: PMC-309 Phase 1a Part B: PMC-309 + Pembrolizumab Phase 1b Cohort A: PMC-309 Phase 1b Cohort B: PMC-309 + Pembrolizumab Estimated overall study duration: approximately 2 to 6 years Dosing Cycle: the duration of a treatment cycle is 3 weeks/21 days.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a participant must meet ALL of the following inclusion criteria:

1. The participant voluntarily signs an informed consent form (ICF) indicating they understand the purpose and procedures required for the study and are willing to participate in the study.
2. Are at least 18 years of age.
3. Are diagnosed with advanced or metastatic solid tumors (non-lymphoma) by histology or pathology that is metastatic or unresectable and considered relapsed and/or refractory to prior therapy.

   Definition of anti-PD-1/L1 refractory participant:

   Participants must have progressed on treatment with an anti-PD1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:
   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   3. PD has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

   i. PD is determined according to iRECIST v1.1. ii. This determination is made by the PI (or designee). Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression
4. Have measurable disease per RECIST v1.1 documented by computerized tomography scan (CT scan) and/or magnetic resonance imaging (MRI), measurable at Baseline. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Have an ECOG performance status of 0 or 1.
6. Can satisfy the following criteria in hematologic, renal, and hepatic function tests performed within 7 days prior to screening:

   1. Hematologic tests:

      * ANC more than and equal to 1.5 × 109 per L.
      * Platelets more than and equal to 100 × 109 per L.
      * Hemoglobin more than and equal to 9.0 g per dL or more than and equal to 5.6 mmol per L.

      Note: Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on a stable dose of erythropoietin (more than equal to approximately 3 months).
   2. Blood coagulation tests:

      * Prothrombin time less than and equal to 1.5 × upper limit of normal (ULN).
      * Activated partial thromboplastin time less than and equal to 1.5 × ULN.
   3. Hepatic function tests:

      * Total bilirubin less than and equal to 1.5 × ULN or direct bilirubin less than and equal to ULN for participants with total bilirubin levels more than and equal to 1.5 × ULN.
      * Aspartate aminotransferase or alanine aminotransferase less than and equal to 2.5 × ULN (less than and equal to 5× ULN in case of liver metastasis).
   4. Renal function test:

      * less than and equal to 1.5 × ULN or creatinine clearance more than and equal to 30 mL/min for participant with creatinine levels above 1.5 × institutional ULN.
7. Are willing and able to adhere to the prohibitions and restrictions as specified in the study protocol.
8. Eligible participants (male and female) of childbearing potential must agree to use reliable contraception (hormone, barrier method, or abstinence) from Screening (Day -1) until at least 120 days after administration of the last dose of the IP.
9. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at Screening (Day -1) and be willing to have additional pregnancy tests as required throughout the study.
10. Human immunodeficiency virus (HIV) infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

    1. Participants on ART must have a CD4+ T-cell count 350 cells/mm3 at time of Screening.
    2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed by HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of Screening and for at least 12 weeks prior to Screening.
    3. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).

Exclusion Criteria:

A participant who meets ANY of the following exclusion criteria must be excluded from the study:

1. Has received treatment with a VISTA targeting agent.
2. Has a history of positive testing for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-hepatitis C virus) or other clinically active liver disease, or positive testing at Screening for HBsAg or anti- hepatitis C virus.
3. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
4. Has a medical condition which, in the opinion of the PI (or designee), places the participant at an unacceptably high risk for toxicity.
5. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
6. Is currently participating in or has participated in a study of an investigational agent or have received anticancer immunotherapy within 4 weeks prior to the first dose of IP.
7. Has an active autoimmune disease with a history of flares requiring immunosuppressant medications within the past 6 months or that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
8. History of known or suspected seizure disorder.
9. Has oxygen-dependent chronic disease.
10. Serious Grade 4 venous thromboembolic event including pulmonary embolism.
11. Participant is receiving therapeutic anticoagulants.
12. Has had an allogeneic tissue/solid organ transplant.
13. Major surgery (eg, requiring general anesthesia) within 4 weeks before the planned first dose of the IP, or not fully recovered from prior surgery, or has surgery planned during the time the participant is expected to participate in the study or within 4 weeks after the last dose of IP.
14. Fertility exclusions:

    1. Participant is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 120 days after the last dose of IP; WOCBP must have a negative pregnancy status confirmed by urine pregnancy test at Screening and within 72 hours of first dose of the IP. (If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.)
    2. Participant is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of the IP.
    3. Male participants must also refrain from sperm donation during the treatment period and for 5 terminal half-lives (of PMC-309) plus an additional 90 days (a spermatogenesis cycle).

    Note: The half-life of PMC-309 is 47 hours.
15. Vaccinated with a live vaccine within 30 days (with the exception of the annual inactivated influenza vaccine) prior to the first dose of the IP.
16. Received COVID-19 vaccine within 7 days of the first IP administration.
17. Any medical condition for which, in the opinion of the PI or designee, participation would not be in the best interest of the participant (eg, compromise the well-being of the participant) or that could prevent, limit, or confound the protocol specified assessments.
18. Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension; poorly controlled diabetes; ongoing active infection requiring antibiotics or acute infectious illness (including suspected viral infection); symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia considered to increase risk for the participant by the PI (or designee); or active psychiatric disorder (schizophrenia, major depressive disorder, bipolar disorder, treated depression with ongoing antidepressant medication etc.) that would limit compliance with study requirements.
19. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (at a dose exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of IP.
20. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, (ie, without evidence of progression for at least 4 weeks by repeat imaging [note that the repeat imaging should be performed during Screening], clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of IP).
21. Prior allogeneic organ or bone marrow transplant.
22. Participant has had prior therapy meeting the following:

    1. Prior T-cell receptor-modified or chimeric antigen receptor T-cell (CART) therapy.
    2. Other anticancer therapy, including chemotherapy, targeted therapy, or treatment with an investigational anticancer agent within 4 weeks prior to the first dose of IP.
    3. Has received prior radiotherapy (excluding limited palliative radiation) within 2 weeks of start of IP or has a history of radiation pneumonitis.
    4. Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (less than and equal to 2 weeks of radiotherapy) to non-CNS disease.
    5. Except for hearing loss, alopecia and pigmentation, all toxicity caused by previous anti-tumor therapy has recovered to Grade 1 or less.
23. Participant received prior therapy with an anti-PD-1 or anti-PD-L1 mAb or with an agent targeting stimulatory or co-inhibitory T-cell receptors and was discontinued from that treatment due to a Grade 3 or higher immune related AE.
24. Participant has an active autoimmune disease that required systemic treatment in the past.
25. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
26. Class III or IV heart failure by New York Heart Association (NYHA) classification.
27. History of abdominal fistula or gastrointestinal perforation within 6 months prior to start of IP administration.
28. History of serious gastrointestinal hemorrhage within 6 months prior to start of IP administration.
29. History of hypertensive crisis or hypertensive encephalopathy.
30. History of posterior reversible encephalopathy syndrome.
31. Social situation that would limit compliance with study requirements.
32. A diagnosis of immunodeficiency or is receiving chronic systemic corticosteroids at a dose that exceeds 10 mg daily of prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior the first dose of the IP. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with abnormal vital signs in response ot treatment with PMC- 309 | Phase 1a and 1b- Upto 35 Cycles (each cycle is 21 days)
  Vital signs will be assessed by changes in systolic/diastolic blood pressure, respiratory rate, body temperature and heart rate.
Number of participants with abnomal clinically significant results with physical examination in response to the treatment with PMC-309 | Phase 1a and 1b- Upto 35 Cycles (each cycle is 21 days)
  A complete physical examinations of general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
Number of participants with abnormal clinically significant 12-lead electrocardiogram (ECG) parameters in response to treatment with PMC-309 | Phase 1a and 1b- Upto 35 Cycles (each cycle is 21 days)
  The following ECG parameters will be recorded: heart rate, RR interval, HR interval, QTc interval, and QRS interval.
Number of participants with abnormal clinically significant laboratory results in response to treatment with PMC-309 | Phase 1a and 1b- Upto 35 Cycles (each cycle is 21 days)
  Laboratory results will include biochemistry, Thyroid function test, hematology, coagulation and urinalysis
Number of participants with adverse events receiving treatment with PMC-309 | Phase 1a and 1b- Upto 35 Cycles (each cycle is 21 days)
  Adverse events includes [treatment-emergent AE, serious AEs, treatment-emergent AEs of special interest] which will be coded using most current version of MedDRA.
Number of participants with abnormal changes in Eastern Cooperative Oncology Group (ECOG) performance status. | Phase 1a and 1b- Screening
Number of participants with abnormal changes in Eastern Cooperative Oncology Group (ECOG) performance status. | Day1 of every cycle (each cycle is 21 days)
To determine the maximum tolerated dose (MTD) of PMC-309 monotherapy (Part A) and establish the preliminary RP2D of PMC-309. | Upto 21 days
  MTD of PMC-309 will be calculated by incidence of DLT at 21 days from the first dosing of PMC 309.
To determine the MTD and establish the preliminary RP2D of PMC-309 when administered in combination with pembrolizumab at 200 mg (Part B). | Upto 21 Days
  MTD of PMC-309 by incidence of DLT at 21 days from the first dosing of PMC-309 in combination with pembrolizumab.

SECONDARY OUTCOMES:
To assess the clinical efficacy of PMC-309 in the treatment of advanced or metastatic solid tumors by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Upto 35 Cycles (each cycle is 21 days)
  RECIST consisting of overall response rate (ORR), disease control rate (DCR) and progression-free survival (PFS) will be graded following CT/MRI of chest, abdomen and pelvis.
The plasma pharmacokinetic endpoints of the study is assessed by peak serum concentration (Cmax) | Upto 35 Cycles (each cycle is 21 Days)
The plasma pharmacokinetic endpoints of the study is assessed by time to peak plasma concentration (Tmax) | Upto 35 Cycles (each cycle is 21 Days)
PK parameter assessed by serum concentration at specified timepoints for area under curve (AUC) | Upto 35 Cycles (each cycle is 21 Days)
To assess the clinical efficacy of PMC-309 at the RP2D as a monotherapy and in combination with pembrolizumab | Upto 35 Cycles (each cycle is 21 Days)
  This will be assessed by RECIST v1.1.
PK parameter assessed by serum concentration over time of PMC-309 at the RP2D as a monotherapy and in combination with pembrolizumab. | Upto 35 Cycles (each cycle is 21 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tazbirkova, Dr, Principal Investigator — Pindara Private Hospital
Locations (4):
- Australia (4):
  - Australian Hospital Care (Pindara) PTY LTD. Trading as Pindara Private Hospital, Benowa, Queensland
  - Ballarat Regional Integrated Cancer Centre (Grampians Health), Ballarat, Victoria
  - Cabrini Health Limited, Malvern, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No